CLINICAL TRIAL: NCT00065182
Title: WEEKLY IV TOPOTECAN/DOCETAXEL COMBINATION COMPARED TO DOCETAXEL IN PATIENTS WITH PRETREATED ADVANCED NSCLC: AN OPEN-LABEL MULTICENTER RANDOMIZED PHASE III TRIAL
Brief Title: Comparison of IV Topotecan/Docetaxel to Docetaxel Alone in Second-Line Stage IIIB/IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104864/615; 2004-002892-17 (EudraCT Number)
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer, Non-Small Cell; Non-Small-Cell Lung Cancer
Keywords: HYCAMTIN; TAXOTERE; non-small cell lung cancer; NSCLC; docetaxel; topotecan; Stage IIIB/IV; Advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Topotecan; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Topotecan/Docetaxel combination
Drug: Docetaxel
  Other Names: Topotecan/Docetaxel combination

SUMMARY:
The purpose of this study is to compare the efficacy and safety of a weekly regimen of two FDA approved drugs in combination versus one FDA approved drug in subjects with advanced non-small cell lung cancer who have received one previous chemotherapy excluding TAXOTERE or HYCAMTIN.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* At least 18 years old
* Confirmed advanced non-small cell lung carcinoma (NSCLC)
* Received one prior chemotherapy for metastatic NSCLC excluding TAXOTERE or HYCAMTIN. In addition, subjects are allowed to have previously received a non-cytotoxic therapy, such as an endothelial growth factor receptor (EGFR) or angiogenesis inhibitor.
* Presence of either measurable or non-measurable disease by radiologic study or physical examination.
* Full recovery and at least 21 days from prior treatment for NSCLC; 42 days from treatment with mitomycin or nitrosureas and 30 days from prior non-cytotoxic therapy.
* At least 3 weeks since last major surgery (a lesser period is acceptable if deemed in the best interest of the patient).
* At least 7 days since prior radiotherapy.
* A probable life expectance of at least 3 months.
* Adequate bone marrow reserve, CBC/Platelet, kidney and liver function.

Exclusion criteria:

* Concomitant malignancies or other malignancies within the last five years.
* Symptoms of brain metastases requiring treatment with steroids.
* Active infection.
* Severe medical problems other than the diagnosis of NSCLC that would limit the ability of the subject to follow study guidelines or expose the subject to extreme risk.
* Ongoing or planned chemotherapy (other than treatment during this study), immunotherapy, radiotherapy, or investigational therapy for the treatment of NSCLC.
* Use of investigational drug within 30 days or 5 half-lives prior to the first dose of study medication.
* Women who are pregnant or lactating.
* Subjects of child-bearing potential refusing to practice adequate contraception.
* Prior treatment with or history of allergic reaction to either HYCAMTIN or TAXOTERE.
* Subjects who cannot receive steroid premedication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2003-08-14 (Actual); Primary Completion 2007-08-30 (Actual); Study Completion 2007-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- United States (62):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Lakeland, Florida
  - GSK Investigational Site, Miami Shores, Florida
  - GSK Investigational Site, Orange Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Decatur, Illinois
  - GSK Investigational Site, Elk Grove Village, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Urbana, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Bowling Green, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Grosse Pointe Woods, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Robbinsdale, Minnesota
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, New Hyde Park, New York
  - GSK Investigational Site, Nyack, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Dunmore, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Hilton Head Island, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Sheboygan, Wisconsin
  - GSK Investigational Site, Casper, Wyoming
- Canada (12):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, St. Catharines, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Weston, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
- Poland (5):
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Szczecin Zdunowo 20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 62 centers: 11 in Canada, 5 in Poland, and 46 in the United States from 14 August 2003 to 30 August 2007. A total of 399 participants with advanced non-small cell lung cancer (NSCLC) were enrolled in the study and randomized to treatment.
Pre-assignment Details: Based on the interim analysis results, the independent data monitoring committee (IDMC) recommended termination of the combination group due to increased toxicity as well as a low likelihood of demonstrating an overall survival benefit at the final analysis.
Groups:
- IV Topotecan + IV Docetaxel: Eligible participants received intravenous (IV) topotecan 3.5 milligrams per square meter per day (mg/m^2/day) and IV docetaxel 30 mg/m^2/day on Days 1, 8 and 15 (± 2 days) of every 28 day treatment cycle. Participants received at least 4 cycles of treatment unless disease progression was noted or the participant withdrew from the study.
- IV Docetaxel: Eligible participants received single-agent IV docetaxel administered either 75 mg/m^2/day Day 1 (± 2 days) of each 21 day treatment cycle or 35 mg/m^2/day on Days 1, 8 and 15 (± 2 days) of each 28 day treatment cycle, based on the investigator's choice. Participants received at least 4 cycles of treatment unless disease progression was noted or the participant withdrew from the study.
Period: Overall Study
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Started | 202 | 197
Completed | 154 | 160
Not Completed | 48 | 37
Not completed — Adverse Event | 24 | 17
Not completed — Lost to Follow-up | 0 | 4
Not completed — Protocol Violation | 3 | 4
Not completed — Serious adverse events (SAE) | 1 | 0
Not completed — Sponsor Decision | 11 | 7
Not completed — Withdrawal by Subject | 8 | 3
Not completed — No clinical benefit | 1 | 0
Not completed — Death | 0 | 1
Not completed — Decline in Status | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- IV Topotecan + IV Docetaxel: Eligible participants received IV topotecan 3.5 mg/m^2/day and IV docetaxel 30 mg/m^2/day on Days 1, 8 and 15 (± 2 days) of every 28 day treatment cycle. Participants received at least 4 cycles of treatment unless disease progression was noted or the participant withdrew from the study.
- IV Docetaxel: Eligible participants received single-agent IV docetaxel administered either 75 mg/m^2/day Day 1 (±2 days) of each 21 day treatment cycle or 35 mg/m^2/day on Days 1, 8 and 15 (± 2 days) of each 28 day treatment cycle, based on the investigator's choice. Participants received at least 4 cycles of treatment unless disease progression was noted or the participant withdrew from the study.
- Total: Total of all reporting groups
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel | Total
Number analyzed (Participants) | 202 | 197 | 399
Age, Customized [Count of Participants; unit: Participants]
  18-40 | 4 | 1 | 5
  41-64 | 129 | 116 | 245
  >=65 | 69 | 80 | 149
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 78 | 141
  Male | 139 | 119 | 258
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 184 | 183 | 367
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Median Time of Overall Survival
Description: Overall survival was defined as the time from randomization to death and it occurs when all randomized participants had at least one year of follow-up past their date of randomization to treatment.
Time Frame: Up to one year from Day -1 (randomization)
Population: Intent-to-treat (ITT) population was defined as all participants randomized to one of the two treatment regimens.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 202 | 197
Weeks | 30.7 [26.1 to 35.9] | 28.6 [23.6 to 36.4]
Statistical Analysis 1: Comparison: IV Topotecan + IV Docetaxel vs IV Docetaxel; Test type: Superiority; p = 0.9460, Log Rank; Hazard Ratio (HR) = 1.007, 95% CI 2-sided [0.813 to 1.248] — Unadjusted hazard ratio
Statistical Analysis 2: Comparison: IV Topotecan + IV Docetaxel vs IV Docetaxel; Test type: Superiority; Hazard Ratio (HR) = 0.977, 95% CI 2-sided [0.788 to 1.210] — Adjusted hazard ratio

2. Secondary Outcome: Number of Participants With One-year Survival
Description: Number of participants with one-year survival were planned to be reported.
Time Frame: Up to one year from Day -1 (randomization)
Population: ITT population. Data was not collected for this outcome measure.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Median Time to Progression
Description: Time to progression is defined as the time between randomization and the first radiologically or clinically documented evidence of progression.
Time Frame: Up to one year from Day -1 (randomization)
Population: ITT population. Data was not collected for this outcome measure.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Response Rate
Description: Response rate is defined as the percentage of participants in the ITT population attaining an overall best response of complete or partial response.
Time Frame: Up to one year from Day -1 (randomization)
Population: ITT population. Data was not collected for this outcome measure.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Response Duration
Description: Response duration is defined as the time from initial radiologically documented response to the first radiologically or clinically documented sign of progression.
Time Frame: Up to one year from Day -1 (randomization)
Population: ITT population. Data was not collected for this outcome measure.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Response-assessed Every 8 Weeks
Description: Time to response is defined as the time between randomization and the first radiologically documented complete or partial response.
Time Frame: Every 8 Weeks post randomization
Population: ITT population. Data was not collected for this outcome measure.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Assessment of Quality of Life-assessed Every 4 Weeks
Description: The effect of treatment regimens on participants-perceived disease status and well-being was assessed using Lung Cancer Symptom Scale (LCSS) that consists of 9 items addressing the time frame of past day: 6 measuring major symptoms for lung malignancies (loss of appetite, fatigue, cough, dyspnea, hemoptysis and pain) and 3 summation items related to total symptomatic distress, activity status and global quality of life. All items are measured by visual analogue scales (VAS) which uses 100 millimeter (mm) lines to determine the intensity of participant responses. The lowest level of symptom intensity or functional disability on the VAS is on left (none) and highest intensity is on right (as much as could be).
Time Frame: Every 4 Weeks post randomization
Population: ITT population. Data was not collected for this outcome measure.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or it is considered to be medically significant.
Time Frame: Up to 16 months
Population: mITT Population was defined as all participants who were randomized and received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 200 | 195
Participants
  Any AEs | 186 | 172
  Any SAEs | 58 | 49

9. Secondary Outcome: Number of Participants With Grade 1, 2, 3 or 4 Hematologic Toxicities
Description: Hematology parameters included hemoglobin, hematocrit, red blood cell count, white blood cell count with differential leukocyte and platelet count. Differential to include total neutrophils, bands, lymphocytes, monocytes, eosinophil, and basophils. Recording of any hematology toxicity grade was done using National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 2.0. Higher the grade, more is the toxicity. Data for number of participants with grade 1, 2, 3 or 4 hematologic toxicities have been presented.
Time Frame: Up to 16 months
Population: mITT population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 200 | 195
Participants
  Hemoglobin, Grade 1: number analyzed (Participants) | 197 | 189
  Hemoglobin, Grade 1 | 76 | 107
  Hemoglobin, Grade 2: number analyzed (Participants) | 197 | 189
  Hemoglobin, Grade 2 | 95 | 46
  Hemoglobin, Grade 3: number analyzed (Participants) | 197 | 189
  Hemoglobin, Grade 3 | 18 | 11
  Neutrophils, Grade 1: number analyzed (Participants) | 197 | 188
  Neutrophils, Grade 1 | 27 | 14
  Neutrophils, Grade 2: number analyzed (Participants) | 197 | 188
  Neutrophils, Grade 2 | 37 | 7
  Neutrophils, Grade 3: number analyzed (Participants) | 197 | 188
  Neutrophils, Grade 3 | 47 | 7
  Neutrophils, Grade 4: number analyzed (Participants) | 197 | 188
  Neutrophils, Grade 4 | 20 | 11
  Platelets, Grade 1: number analyzed (Participants) | 197 | 188
  Platelets, Grade 1 | 75 | 10
  Platelets, Grade 2: number analyzed (Participants) | 197 | 188
  Platelets, Grade 2 | 20 | 3
  Platelets, Grade 3: number analyzed (Participants) | 197 | 188
  Platelets, Grade 3 | 18 | 0
  Platelets, Grade 4: number analyzed (Participants) | 197 | 188
  Platelets, Grade 4 | 1 | 0
  White blood cell, Grade 1: number analyzed (Participants) | 197 | 189
  White blood cell, Grade 1 | 38 | 28
  White blood cell, Grade 2: number analyzed (Participants) | 197 | 189
  White blood cell, Grade 2 | 51 | 14
  White blood cell, Grade 3: number analyzed (Participants) | 197 | 189
  White blood cell, Grade 3 | 50 | 13
  White blood cell, Grade 4: number analyzed (Participants) | 197 | 189
  White blood cell, Grade 4 | 15 | 2

10. Secondary Outcome: Number of Participants With Grade 3 or 4 Clinical Chemical Toxicities
Description: Standard chemistry evaluation included sodium, potassium, chloride, bicarbonate, calcium, phosphorous, magnesium, blood urea nitrogen (BUN)/urea, uric acid, creatinine, lactate dehydrogenase (LDH), aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin, total protein and albumin. Recording of any hematology toxicity grade was done using National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 2.0. Higher the grade, more is the toxicity. Data for number of participants with grade 3 or 4 clinical chemical toxicities have been presented.
Time Frame: Up to 16 months
Population: mITT population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 200 | 195
Participants
  Albumin, Grade 3: number analyzed (Participants) | 177 | 182
  Albumin, Grade 3 | 3 | 3
  BUN/Urea, Grade 3: number analyzed (Participants) | 187 | 191
  BUN/Urea, Grade 3 | 4 | 2
  Creatinine, Grade 3: number analyzed (Participants) | 185 | 186
  Creatinine, Grade 3 | 0 | 1
  Alkaline Phosphatase, Grade 3: number analyzed (Participants) | 180 | 181
  Alkaline Phosphatase, Grade 3 | 1 | 1
  AST, Grade 3: number analyzed (Participants) | 182 | 185
  AST, Grade 3 | 0 | 1
  AST, Grade 4: number analyzed (Participants) | 82 | 185
  AST, Grade 4 | 1 | 0
  ALT, Grade 3: number analyzed (Participants) | 183 | 185
  ALT, Grade 3 | 1 | 0
  ALT, Grade 4: number analyzed (Participants) | 183 | 185
  ALT, Grade 4 | 1 | 0
  Bilirubin, Grade 3: number analyzed (Participants) | 182 | 183
  Bilirubin, Grade 3 | 1 | 2
  Sodium, Grade 3: number analyzed (Participants) | 184 | 187
  Sodium, Grade 3 | 12 | 9
  Sodium, Grade 4: number analyzed (Participants) | 184 | 187
  Sodium, Grade 4 | 0 | 1
  Calcium, Grade 3: number analyzed (Participants) | 180 | 182
  Calcium, Grade 3 | 2 | 2
  Calcium, Grade 4: number analyzed (Participants) | 180 | 182
  Calcium, Grade 4 | 0 | 1
  Potassium, Grade 3: number analyzed (Participants) | 185 | 187
  Potassium, Grade 3 | 7 | 3
  Potassium, Grade 4: number analyzed (Participants) | 185 | 187
  Potassium, Grade 4 | 1 | 1
  Magnesium, Grade 3: number analyzed (Participants) | 167 | 171
  Magnesium, Grade 3 | 4 | 2

11. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs Data
Description: Vital sign parameters included (blood pressure, and pulse rate after five minutes sitting, body temperature). Blood pressure and pulse rate was measured after sitting for 5 minutes. Only participants with clinically significant abnormal Vital sign data was reported.
Time Frame: Up to 16 months
Population: mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
Number analyzed (Participants) | 200 | 195
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 16 months
Description: mITT population was analyzed for safety data.
Arm/Group | IV Topotecan + IV Docetaxel | IV Docetaxel
All-Cause Mortality (participants affected / at risk) | 170/200 | 165/195
Serious Adverse Events (participants affected / at risk) | 58/200 | 49/195
Other Adverse Events (participants affected / at risk) | 181/200 | 166/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IV Topotecan + IV Docetaxel (N=200) | IV Docetaxel (N=195)
Pneumonia (Infections and infestations) | 7 | 4
Anaemia (Blood and lymphatic system disorders) | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Catheter related complication (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Electrocardiogram ST-T change (Investigations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Infusion site phlebitis (General disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Shock (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Perforated ulcer (Gastrointestinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Topotecan + IV Docetaxel (N=200) | IV Docetaxel (N=195)
Fatigue (General disorders) | 90 | 74
Oedema peripheral (General disorders) | 28 | 31
Pyrexia (General disorders) | 31 | 28
Asthenia (General disorders) | 19 | 21
Chest pain (General disorders) | 17 | 19
Oedema (General disorders) | 8 | 10
Mucosal inflammation (General disorders) | 11 | 6
Nausea (Gastrointestinal disorders) | 57 | 43
Diarrhoea (Gastrointestinal disorders) | 51 | 40
Constipation (Gastrointestinal disorders) | 39 | 38
Vomiting (Gastrointestinal disorders) | 26 | 22
Abdominal pain (Gastrointestinal disorders) | 12 | 11
Stomatitis (Gastrointestinal disorders) | 12 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 29
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 15 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Headache (Nervous system disorders) | 24 | 20
Dysgeusia (Nervous system disorders) | 13 | 20
Dizziness (Nervous system disorders) | 21 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 12 | 7
Neuropathy peripheral (Nervous system disorders) | 8 | 10
Anaemia (Blood and lymphatic system disorders) | 44 | 21
Neutropenia (Blood and lymphatic system disorders) | 34 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 2
Anorexia (Metabolism and nutrition disorders) | 33 | 37
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 8
Dehydration (Metabolism and nutrition disorders) | 10 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 36 | 35
Rash (Skin and subcutaneous tissue disorders) | 10 | 18
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 17
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Insomnia (Psychiatric disorders) | 19 | 28
Anxiety (Psychiatric disorders) | 11 | 11
Confusional state (Psychiatric disorders) | 10 | 3
Lacrimation increased (Eye disorders) | 5 | 13
Hypotension (Vascular disorders) | 10 | 7

LIMITATIONS AND CAVEATS:
The combination group was terminated as per recommendation of IDMC based on the interim analysis results occurred on 04-November-2005. Therefore all the efficacy parameters were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.